CLINICAL TRIAL: NCT00336492
Title: A Phase 3, Randomized, Open-label, Parallel-group, Multicenter Trial to Evaluate the Safety and Efficacy of Infliximab (REMICADE�) in Pediatric Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of the Safety and Efficacy of Infliximab(REMICADE ) in Pediatric Patients With Moderately to SeverelyActive Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012388; C0168T72 (Other: Centocor)
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; inflammatory bowel disease; children
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Infliximab

ARMS (2):
- 002 (Experimental): infliximab infusion of 5mg/kg at weeks 0, 2, 6 followed by every 12 wks through week 42; infliximab - Could receive infusion of 10mg/kg every 8 weeks up to week 42; infliximab - Could receive infusion of 5mg/kg every 8 weeks up to week 42
  Interventions: Biological: infliximab
- 001 (Experimental): infliximab infusion of 5mg/kg at weeks 0, 2, 6 followed by every 8 wks through week 46; infliximab - Could receive infusion of 10mg/kg every 8 weeks up to week 46
  Interventions: Biological: infliximab

INTERVENTIONS:
Biological: infliximab — infusion of 5mg/kg at weeks 0, 2, 6 followed by every 12 wks through week 42; infliximab - Could receive infusion of 10mg/kg every 8 weeks up to week 42; infliximab - Could receive infusion of 5mg/kg every 8 weeks up to week 42
  Arms: 002
Biological: infliximab — infusion of 5mg/kg at weeks 0, 2, 6 followed by every 8 wks through week 46; infliximab - Could receive infusion of 10mg/kg every 8 weeks up to week 46
  Arms: 001
Biological: infliximab — infliximab - Could receive infusion of 10 mg/kg every 8 weeks up to week 42
  Arms: 002
Biological: infliximab — infusion of 5mg/kg at weeks 0, 2, 6, then every 12 wks through week 42
  Arms: 001

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of infliximab (Remicade) in children with moderately to severely active ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative Colitis (UC) is a disorder involving the lining of the colon. A substance called "tumor necrosis factor" (TNF) naturally occurs in the body. TNF is thought to play an important role in the development of ulcerative colitis by causing some of the damage that is seen in the colon. "Antibodies" are normally made in the body and help fight off infection. Infliximab is an antibody that is made in a scientific laboratory, using parts of both mouse and human antibodies. It has been designed to attach to TNF, making it difficult for TNF to do any damage. This study will be done at centers in North America and Europe. Each child will first have a clinic visit (screening visit) to have some tests done to make sure the child is the type of patient who should be in this study. At the 2nd visit (week 0), the child will have the first treatment with infliximab. All children in the study will receive 5 mg/kg infliximab 3 times (at weeks 0, 2 and 6) over the first 6 weeks of the study. If the child's symptoms do not improve by the 8th week, the child will receive no further infusions, but will return for safety evaluations. If the child's symptoms do improve, the child will be randomly assigned (like the flip of a coin) to either 5 mg/kg infliximab every 8 weeks through week 46 or 5 mg/kg infliximab every 12 weeks through week 42. If the child gets worse after being randomly assigned, the amount of infliximab may be increased or the infliximab may be given more frequently. A final infusion will be given at either week 42 or week 46. There will be a safety evaluation at week 54 and a visit at week 62 to get a blood sample. Patients will receive 5 mg/kg of infliximab at weeks 0, 2 and 6 and then 5mg/kg infliximab either every 8 weeks or 12 weeks until weeks 42 or 46. Infliximab is given as an intravenous infusion over 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Have moderately to severely active ulcerative colitis
* Diagnosed with ulcerative colitis for 2 weeks before screening
* Male patients who are sexually active and female patients who are sexually active or of childbearing potential must use adequate birth control while participation in the study and for 6 months after the last infusion.

Exclusion Criteria:

* History of latent or active TB
* Have had a live viral or bacterial vaccination within 3 months before screening
* Have or have had serious infections within 3 months before screening
* Prior treatment with infliximab

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (27):
- United States (18):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Rochester, Minnesota
  - New Hyde Park, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Providence, Rhode Island
  - Milwaukee, Wisconsin
- Belgium (2):
  - Antwerp
  - Leuven
- Canada (5):
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Toronto, Ontario
  - Edmonton
  - Halifax
- Hvidovre, Denmark
- Rotterdam, Netherlands

REFERENCES:
- [Derived] Singh S, Proudfoot JA, Dulai PS, Jairath V, Fumery M, Xu R, Feagan BG, Sandborn WJ. No Benefit of Concomitant 5-Aminosalicylates in Patients With Ulcerative Colitis Escalated to Biologic Therapy: Pooled Analysis of Individual Participant Data From Clinical Trials. Am J Gastroenterol. 2018 Aug;113(8):1197-1205. doi: 10.1038/s41395-018-0144-2. Epub 2018 Jun 21. PMID 29925913
- See also: A Study of the Safety and Efficacy of Infliximab(REMICADE ) in Pediatric Subjects with Moderately to SeverelyActive Ulcerative Colitis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=174&filename=CR012388_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized Group: Participants who were not randomized at Week 8
- 5 mg/kg Infliximab Every 8 Wks: Participants who were clinical responders at Week 8 who were randomized to 5 mg/kg Infliximab every 8 wks
- 5 mg/kg Infliximab Every 12 Wks: Participants who were clinical responders at Week 8 who were randomized to 5 mg/kg Infliximab every 12 wks
Period: Overall Study
Arm/Group | Not Randomized Group | 5 mg/kg Infliximab Every 8 Wks | 5 mg/kg Infliximab Every 12 Wks
Started | 15 | 22 | 23
Completed | 0 | 18 | 12
Not Completed | 15 | 4 | 11
Not completed — Adverse Event | 4 | 3 | 6
Not completed — Lack of Efficacy | 6 | 1 | 4
Not completed — Other | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Not Randomized Group | 5 mg/kg Infliximab Every 8 Wks | 5 mg/kg Infliximab Every 12 Wks | Total
Number analyzed (Participants) | 15 | 22 | 23 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 11.9 (2.64) | 13.7 (3.20) | 14.2 (3.03) | 13.4 (3.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 13 | 32
  Male | 8 | 10 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Clinical Response at Week 8
Description: Range is 0 to 12 points, where 0 is the least disease activity, and 12 is the most disease activity. Clinical response at Week 8 is defined as a decrease from baseline in the Mayo score(based on symptoms of ulcerative colitis) by >=30% and >= 3 points, with a decrease in the rectal bleeding subscore >=1 or a rectal bleeding subscore of 0 or 1. Treatment failure rules (patients who discontinued study agent due to lack of therapeutic effect, had a colectomy or ostomy, or had protocol-prohibited medication changes) were applied to determine the final clinical response status for each patient.
Time Frame: Week 8
Population: The primary efficacy endpoint analysis was based on all treated participants.
Measure: Number; unit: Participants
Groups:
- Infliximab 5 mg/kg: Infliximab 5 mg/kg group
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 60
Participants | 44

2. Secondary Outcome: The Number of Participants With Pediatric Ulcerative Colitis Activity Index (PUCAI) Remission at Week 54
Description: Range is 0 to 85 points, where 0 is the least disease activity, and 85 is the most disease activity. Remission is a score <10. In addition to the PUCAI remission status, treatment failure rules (patients who discontinued study agent due to lack of therapeutic effect, had a colectomy or ostomy, had protocol-prohibited medication changes, or stepped up) were applied to determine the final PUCAI.
Time Frame: Week 54
Population: PUCAI remission at Week 54 analysis was based on all participants randomized at Week 8 who were evaluable for PUCAI. Fifteen participants discontinued Infliximab treatment.
Measure: Number; unit: Participants
Arm/Group | 5 mg/kg Infliximab Every 8 Wks | 5 mg/kg Infliximab Every 12 Wks
Number analyzed (Participants) | 21 | 22
Participants | 8 | 4
Statistical Analysis 1: Comparison: 5 mg/kg Infliximab Every 8 Wks vs 5 mg/kg Infliximab Every 12 Wks; Test type: Superiority or Other; p = 0.146, Chi-squared

ADVERSE EVENTS:
Description: Data for subjects who stepped up are included according to the regimen received before step-up.
Arm/Group | Not Randomized Group | 5 mg/kg Infliximab Every 8 Wks | 5 mg/kg Infliximab Every 12 Wks
Serious Adverse Events (participants affected / at risk) | 5/15 | 4/22 | 5/23
Other Adverse Events (participants affected / at risk) | 10/15 | 19/22 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Not Randomized Group (N=15) | 5 mg/kg Infliximab Every 8 Wks (N=22) | 5 mg/kg Infliximab Every 12 Wks (N=23)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 4 | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Infection Viral (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 0 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia Lobar (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Not Randomized Group (N=15) | 5 mg/kg Infliximab Every 8 Wks (N=22) | 5 mg/kg Infliximab Every 12 Wks (N=23)
Anemia (Blood and lymphatic system disorders) | 0 | 4 | 2
Thrombocythemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 3 | 3 | 2
Blood in Stool (Gastrointestinal disorders) | 1 | 0 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 7 | 15
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Stomatitis Ulcerative (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Chest Pain (General disorders) | 1 | 0 | 1
Chills (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 4
Hepatic Enzymes Increased (Hepatobiliary disorders) | 0 | 0 | 2
Fever (Infections and infestations) | 1 | 6 | 1
Infection Bacterial (Infections and infestations) | 1 | 0 | 0
Inflammation (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 2
Influenza-Like Symptoms (Infections and infestations) | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 3
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Thinking Abnormal (Psychiatric disorders) | 1 | 0 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Hemorrhoids (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days